CLINICAL TRIAL: NCT05843396
Title: Brain Organization, Development, and Response to Intervention in Individual Neonates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1368060
Record Dates: First submitted 2023-01-23; First posted 2023-05-06 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Development, Infant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neonatal Massage Received (Active Comparator)
  Interventions: Behavioral: Neonatal Massage
- No Massage Received (No Intervention)

INTERVENTIONS:
Behavioral: Neonatal Massage — caregivers providing therapeutic touch techniques on their neonate
  Arms: Neonatal Massage Received

SUMMARY:
The goal of this study is to learn about brain connectivity and if massaging babies shortly after birth has an impact. Half of the recruited babies will receive massage daily while the other half will not, and differences will be observed.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Ability to give informed consent

Exclusion Criteria:

* Prisoners (vulnerable population)
* Pregnant women <18 years of age
* Active psychosis, mania, suicidal ideation (safety)
* Active substance dependence
* Non-singleton pregnancy (e.g., twins)
* Gestational Age <36 weeks (neonates)
* Neonatal encephalopathy (neonates)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Change in correlated brain activity among functional brain areas in the somatomotor cortex | up to 3 months
  Brain activity is measured across the brain with functional magnetic resonance imaging (fMRI) before and after the intervention. The timeseries of brain activity will be extracted from each of the subject-specific parcels of the somatomotor network (SMN). Parcels will be divided into those that represent the upper versus lower extremity. The average of the pairwise correlations in the timeseries between upper and lower extremity parcels is the "cross-effector SMN functional connectivity" that is the primary measure. This measure will be computed before and after the intervention; we predict a decrease in cross-effector SMN functional connectivity following the intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Undecided